CLINICAL TRIAL: NCT05620342
Title: Administration of T Cells Expressing a 2nd Generation GD2 Chimeric Antigen Receptor, IL-15, and iCaspase9 Safety Switch in Subjects With Lung Cancer
Brief Title: Autologous CAR T-Cells Targeting the GD2 Antigen for Lung Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry); United States Department of Defense (U.S. Federal Agency); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2115-ATL
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Small Cell Lung Carcinoma; Non Small Cell Lung Cancer
Keywords: cellular therapy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iC9.GD2.CAR.IL-15 T Therapy (Experimental): Experimental: Single Arm Subjects with extensive stage lung cancer or stage IV non-small cell lung cancer that is platinum-refractory and received PD-1 and/or PD-L1 therapy will receive iC9.GD2.CAR.IL-15 T cells were manufactured from their collected blood sample.
  Interventions: Biological: iC9.GD2.CAR.IL-15 T Infusion

INTERVENTIONS:
Biological: iC9.GD2.CAR.IL-15 T Infusion — iC9-GD2.CAR.IL-15 T-cells product will be administered via intravenous injection over 5 - 10 minutes.

SUMMARY:
This is a phase 1, single-center, open-label study that enrolls adult subjects with extensive stage lung cancer or stage IV non-small cell lung cancer that is platinum-refractory and received PD-1 and/or PD-L1 therapy. The purpose of this study is to test the safety of using a new treatment called autologous T lymphocyte chimeric antigen receptor cells against the GD2 antigen (iC9-GD2.CAR.IL-15 T cells) in subjects with lung cancer. How much (dose) of the iC9-GD2.CAR.IL-15 T cells are safe to use without causing too many side effects and what is the maximum dose that could be tolerated will be studied.

Modified immune cells as an experimental treatment that combines antibodies and T cells will be used. Antibodies are proteins that protect the body from foreign invaders like bacteria. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill viruses and other cells, including tumor cells. Although antibodies and T cells have been used to treat cancer and they both have shown promise, neither alone has been able to cure most patients. This study will combine T cells and antibodies to create a more effective treatment.

The treatment that is being researched in this study is called autologous T lymphocyte chimeric antigen receptor cells targeted against the disialoganglioside (GD2) antigen that expresses Interleukin (IL)-15, and the inducible caspase 9 safety switch (iC9). The short name for this treatment is iC9.GD2.CAR.IL-15 T cells therapy is an experimental therapy and has not been approved by the Food and Drug Administration. There are two steps. In the first step, blood will be collected from the subjects to prepare the iC9-GD2.CAR.IL-15 T cells. T cells will be isolated from the blood and modified to make iC9-GD2.CAR.IL-15. In the second step, the iC9-GD2.CAR.IL-15 T cells produced from the subject's own blood will be administered to the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to undergo cell procurement explained to, understood by, and signed by the subject.
2. Subject has a life expectancy of ≥ 12 weeks.
3. Subject must be platinum-refractory and either currently receiving or has previously received a PD1/PDL1 inhibitor
4. Use of systemic corticosteroids at doses ≥10 mg prednisone daily or it's equivalent; those receiving <10 mg daily may be enrolled at the discretion of the investigator.
5. Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to cell procurement.
6. Subject has demonstrated adequate organ function.

Exclusion Criteria:

1 . Subject has less than 12 weeks of life expectancy.

2. Subject did not receive platinum-based chemotherapy

3. Subject does not have adequate organ function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2027-11-24 (Estimated); Study Completion 2029-10-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse event | Up to 4 weeks
  The number of participants with adverse events (AE)s will be reported as a measure of the safety and tolerability of C9.GD2.CAR.IL-15 T. AEs will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Cytokine Release Syndrome (CRS) | Up to 4 weeks
  CRS will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading.
  Grade 1 - Mild (Symptomatic Management): Fever ≥38^ o C, No hypotension, No hypoxia, Grade 2 - Moderate (Moderate Intervention): Fever ≥38^ o C, Hypotension not requiring vasopressors, Hypoxia requiring low-flow nasal cannula (≤6 L/minute) or blow-by, Grade 3 - Severe (Aggressive Intervention): Fever ≥ 38^ o C , Hypotension requiring a vasopressor with or without vasopressin, Hypoxia requiring high-flow nasal cannula (>6 L/minute), facemask, nonrebreather mask, or Venturi mask, Grade 4 - Life-threatening (Life-sustaining intervention): Fever ≥38^oC, Hypotension requiring multiple vasopressors (excluding vasopressin), Hypoxia requiring positive pressure (e.g. Continuous positive airway pressure, BiPAP, intubation, mechanical ventilation), Grade 5 - Death: Death.
Neurotoxicity | Up to 4 weeks
  Neurotoxicity will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) Immune effector cell-associated neurotoxicity syndrome (ICANS) Consensus Grading criteria.
  ICANS grading criteria are outlined in the protocol on a scale from 1 (mild) to 4 (critical) based on the Immune Effector Cell-Associated Encephalopathy (ICE) Score. Grade 1:Score: 7-9 (mild impairment), Grade 2:Score: 3-6 (moderate impairment), Grade 3: Score: 0-2 (severe impairment), Grade 4: Score: Subject in critical condition, and/or obtunded and cannot perform an assessment of tasks.

SECONDARY OUTCOMES:
Identification of Recommended phase 2 dose (RP2D) | Up to 4 weeks
  The RP2D of iC9-GD2.CAR.IL-15 T-cells will be determined based on the modified 3+3 dose-finding rule based on the protocol. Dose escalation will be performed considering the dose-limiting toxicities (DLTs), dose level (DL) will be increased unless there is no DLT.
Overall Response Rate (ORR) | Up to 4 weeks
  ORR will be assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) which defines Complete Response (CR) as the disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall Response Rate (ORR) = number of subjects who achieved CR + number of subjects who achieved PR / total number of subjects who received the study treatment.
Progression Free Survival (PFS) | Up to 2 years
  PFS will be measured from the first day of lymphodepletion chemotherapy prior to iC9-GD2.CAR.IL-15 T-cell infusion to progression based on RECIST 1.1 criteria or death.
  RECIST 1.1 Criteria: Stable Disease (SD): No response or less response than Partial or Progressive and Progressive Disease (PD): A 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall Survival (OS) | Up to 2 years
  OS will be measured from the first day of lymphodepletion chemotherapy prior to iC9-GD2.CAR.IL-15 T-cell infusion to date of death for any cause.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from documentation of partial response or response to disease progression based on RECIST 1.1.
  RECIST 1.1 Criteria: Complete Response (CR) as the disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall Response Rate (ORR) = number of subjects who achieved CR + number of subjects who achieved PR / total number of subjects who received the study treatment.Stable Disease (SD): No response or less response than Partial or Progressive and Progressive Disease (PD): A 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Duration of Benefit | Up to 2 years
  Duration of benefit is defined as the time from the first day of lymphodepletion chemotherapy prior to iC9-GD2.CAR.IL-15 T-cell infusion to disease progression, next therapy, or death.
  RECIST 1.1 Criteria Progressive Disease (PD): A 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Disialoganglioside (GD2) Expression | Baseline
  GD2 Expression will be measured via immunohistochemistry (IHC) on tumor samples collected from subjects.
Disialoganglioside Expression and tumor response rate correlations | Up to 2 years
  GD2 value and tumor response rate graded according to RECIST 1.1 relation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, Principal Investigator — jared_weiss@med.unc.edu
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials